CLINICAL TRIAL: NCT06532032
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of Amivantamab and Docetaxel Combination Therapy in Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Combination Therapy With Amivantamab and Docetaxel in Participants With Metastatic Non-small Cell Lung Cancer
Acronym: swalloWTail
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 61186372PANSC2003; 61186372PANSC2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Combination Dose Selection) (Experimental): Participants will receive amivantamab intravenous (IV) infusion administered based on body weight from Cycle 1 Day 1, Day 2, and subsequent doses on Days 8 and 15, and then on Day 1 of each 21-day treatment cycle. Docetaxel will be administered on Day 2 of Cycle 1 (before Day 2 amivantamab infusion) and then on Day 1 of each 21-day treatment cycle, thereafter. Doses will be escalated or de-escalated based on the dose limiting toxicities (DLTs) and the recommended Phase 2 combination dose (RP2CD) will be determined. Participants will continue study treatment until disease progression, unacceptable toxicity, or until another criterion for discontinuation of study treatment is met.
  Interventions: Drug: Amivantamab; Drug: Docetaxel
- Phase 2 (Dose Expansion) (Experimental): Participants will receive amivantamab in combination with docetaxel in 2 cohorts (Cohort A [adenocarcinoma] and Cohort B [squamous]) at the RP2CD determined in Phase 1. Participants will continue study treatment until disease progression, unacceptable toxicity, or until another criterion for discontinuation of study treatment is met.
  Interventions: Drug: Amivantamab; Drug: Docetaxel

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered as IV infusion.
  Other Names: JNJ-61186372
Drug: Docetaxel — Docetaxel will be administered as IV infusion.
  Other Names: TAXOTERE

SUMMARY:
The purpose of this study is to identify the recommended Phase 2 (combination) dose (RP2CD) of the amivantamab and docetaxel combination therapy in participants with metastatic non-small cell lung cancer (NSCLC) in Phase 1 (combination dose selection); and to evaluate the antitumor effect of the combination at the selected RP2CD in participants with NSCLC without oncogenic driver mutations with disease progression on platinum-based chemotherapy and immune checkpoint inhibitor, in the Phase 2 (expansion).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed NSCLC and must have metastatic NSCLC at the time of enrollment
* Participant must have at least 1 measurable lesion, according to RECIST v1.1, that has not been previously irradiated
* May have brain metastases only if previously definitively treated, and participant is clinically stable and asymptomatic for >2 weeks and is off or receiving low-dose corticosteroid treatment (<=10 mg prednisone or equivalent) for at least 2 weeks prior to start of study treatment
* May have a prior malignancy (other than the disease under study) if the natural history or treatment is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Have an ECOG performance status of 0 or 1

Exclusion Criteria:

* For Phase 2 only: Participant has known oncogenic driver mutations (EGFR, MET, HER2, ALK, ROS1, NTRK, BRAF, RET, or KRAS) as detected by local testing or by central ctDNA testing
* Participant has received radiotherapy for palliative purposes less than 14 days prior to the first dose of study treatment
* Participant has: a.(Or has a history of) leptomeningeal disease (carcinomatous meningitis); b. Spinal cord compression not definitively treated with surgery or radiation.
* Medical history of (non-infectious) ILD/pneumonitis, or has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening- Participant has history of any significant drug allergy (such as anaphylaxis, hepatotoxicity, or immune-mediated thrombocytopenia or anemia) or has known allergies, hypersensitivity, or intolerance to: a. amivantamab or amivantamab excipients (refer to the amivantamab IB); b.docetaxel, docetaxel excipients or to other drugs formulated with polysorbate and paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse events (AEs) by Severity | Up to 1 year 4 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 1: Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 21 days
  DLTs are specific adverse events and are defined as any of following: Any high grade (Grade 3, 4 or 5) non-hematologic toxicity with exceptions such as: Grade 3 fever resolved in <=48 hours, anorexia; Grade 3 nausea, vomiting or diarrhea, or constipation Grade 3 fatigue; rash that improves to Grade <; transient electrolyte abnormalities; symptoms of IRRs that are attributable to amivantamab or docetaxel; Tumor flare; hematologic toxicity (Grade 4 anemia or neutropenia, Febrile neutropenia; Grade 3 or 4 thrombocytopenia associated with bleeding or requiring transfusion); pulmonary toxicity (confirmed any grade pulmonary toxicity, including pneumonitis or interstitial lung disease [ILD]), liver enzyme elevation (ALT or AST elevation>=Grade 3 persisting >=7 days); or treatment delay greater than (>) 28 days due to unresolved toxicity.
Phase 2: Objective Response Rate (ORR) | Up to 1 year 4 months
  ORR is defined as the percentage of participants who achieve either a confirmed partial response (PR) or complete response (CR), using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Number of Participants with AEs by Severity | Up to 1 year 4 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. Severity will be graded according to the NCI-CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 1 and Phase 2: Number of Participants with Abnormalities in Clinical Laboratory Parameters | Up to 1 year 4 months
  Number of participants with abnormalities in clinical laboratory parameters (serum chemistry, hematology, coagulation, serology, and urinalysis) will be reported.
Phase 2 : Duration of Response (DoR) | Up to 1 year 4 months
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death from any case, whichever comes first, for participants who have PR or CR.
Phase 2: Disease Control Rate (DCR) | Up to 1 year 4 months
  DCR is defined as the percentage of participants who achieve a PR, CR, or stable disease using RECIST version 1.1.
Phase 2: Progression Free Survival (PFS) | Up to 1 year 4 months
  PFS is defined as the time from first dose date until the date of disease progression or death, whichever comes first, based on investigator assessment using RECIST version 1.1.
Phase 2: Overall Survival (OS) | Up to 1 year 4 months
  OS is defined as the time from the date of administration of the first study treatment until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research &Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (15):
- United States (6):
  - UCI Health Irvine Hospital, Irvine, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - University of California Irvine Medical Center Chao Family Comprehensive Cancer Center, Orange, California
  - Oncology Hematology Associates, Springfield, Missouri
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Virginia Cancer Specialists, Fairfax, Virginia
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chi Mei Medical Center Liu Ying, Liou Ying Township
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University, Taipei
- Ankara Bilkent Sehir Hastanesi, Çankaya, Turkey (Türkiye)
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Royal Marsden NHS Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency